CLINICAL TRIAL: NCT05434728
Title: Disordered Bleeding in Ehlers Danlos Syndromes
Brief Title: Characterization of Bleeding Disorders in EDS
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Principal Investigator, Nimish Mittal, Medical Director - GoodHope EDS Clinic, Toronto General Hospital, University Health Network, Toronto
Other Study IDs: 21-5787.0
Record Dates: First submitted 2022-06-17; First posted 2022-06-28 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Ehlers-Danlos Syndrome; EDS; Classical Ehlers-Danlos Syndrome; Classical EDS (cEDS); Hypermobile Ehlers-Danlos Syndrome; Hypermobile EDS (hEDS); Vascular Ehlers-Danlos Syndrome; Vascular EDS (vEDS)
MeSH Terms: conditions — Ehlers-Danlos Syndrome; Ehlers-Danlos syndrome type 1; Ehlers-Danlos syndrome type 3; Ehlers-Danlos Syndrome, Type IV

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Venous blood sample will be collected
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Hypermobile EDS: Individuals with a confirmed diagnosis of hypermobile EDS
  Interventions: Other: 20 ml venous blood collection
- Classical EDS: Individuals with a confirmed diagnosis of classical EDS
  Interventions: Other: 20 ml venous blood collection
- Vascular EDS: Individuals with a confirmed diagnosis of vascular EDS
  Interventions: Other: 20 ml venous blood collection

INTERVENTIONS:
Other: 20 ml venous blood collection — participant blood sample will be divided between sample EDTA sample tubes for thrombin generation testing and viscoelastic (ROTEM) testing of impaired hemostasis

SUMMARY:
Ehlers-Danlos Syndrome (EDS) is a disease that weakens the connective tissues (i.e. tendons and ligaments) in the human body. EDS can make the joints loose and alter skin and wound healing. It can also weaken blood vessels and organs. Many EDS patients are referred for investigation of bleeding symptoms. Although most patients will have mild symptoms such as bruising, many will experience significant bleeding that can be life-threatening. The physiological reason behind this has not been identified and therefore, treating this is challenging. In addition, patients with EDS frequently require major surgery due to complications from their connective tissue disease. These surgery carries a significant risk of catastrophic bleeding which is further magnified in this group of patients. The specific reason of clinical bleeding in patients with EDS is likely multifactorial, including skin and blood vessel fragility leading to increased bruising and poor wound healing, coagulopathies related to factor deficiency, acquired vonWillebrand disease (VWD), and notable platelet dysfunction.

Despite compelling preliminary evidence, there is limited data on the diagnosis and management of platelet dysfunction in EDS patients. Therefore, in this study we will characterize hemostasis, the medical term which refers to the process of stopping blood flow, across the three most common subtypes of EDS.we will also determine the burden of illness of pathologic bleeding in patients with Ehlers-Danlos Syndrome (EDS) using validated patient reported tools.

ELIGIBILITY:
Inclusion Criteria:

* Any adult (≥ 18 years) patient with a known diagnosis of Ehlers Danlos Syndrome (Subtypes Classical, Hypermobile, or Vascular) as per the 2017 International Classification of Ehlers Danlos Syndrome.

Exclusion Criteria:

* Subtypes of Ehlers Danlos Syndrome which are not Classical, Hypermobile, or Vascular.
* Unable or unwilling to consent for the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Any adult (≥ 18 years) patient with a known diagnosis of Ehlers Danlos Syndrome (Subtypes Classical, Hypermobile, or Vascular) as per the 2017 International Classification of Ehlers Danlos Syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
The prevalence of platelet dysfunction among patients with a known diagnosis of EDS | 6 months

SECONDARY OUTCOMES:
The severity of platelet dysfunction (as characterized by the percentage of non-functional platelets) in patients with EDS | 6 months
The prevalence and severity of impaired thrombin generation as assessed through thrombin generation testing in patients with EDS | 6 months
The prevalence and severity of impaired hemostasis as assessed through viscoelastic testing (ROTEM) in patients with EDS | 6 months
The prevalence and severity of bleeding as assessed via the ISTH-BAT scale in patients with EDS | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Nimish Mittal, MBBS, MD, Principal Investigator — University Health Network - University of Toronto
Locations (1):
- GoodHope EDS - Toronto General Hospital, Toronto, Ontario, Canada